CLINICAL TRIAL: NCT00041210
Title: Protocol for a Randomized Phase III Study of the Stanford V Regimen, Compared With ABVD for the Treatment of Advanced Hodgkin's Disease
Brief Title: Combination Chemotherapy in Treating Patients With Previously Untreated Advanced Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mount Vernon Cancer Centre at Mount Vernon Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069453; BNLI-STANFORDV; EU-20206
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-04

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; ABVD protocol; Dacarbazine; Doxorubicin; Etoposide; Mechlorethamine; Prednisone; Vinblastine; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: ABVD regimen
Drug: Stanford V regimen
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: mechlorethamine hydrochloride
Drug: prednisone
Drug: vinblastine sulfate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating patients who have advanced Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different combination chemotherapy regimens in treating patients who have advanced Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare relapse-free and overall survival of patients with previously untreated advanced Hodgkin's lymphoma treated with bleomycin, doxorubicin, etoposide, mechlorethamine, vinblastine, vincristine, and prednisone (Stanford V) vs doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD).
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (Stanford V): Patients receive mechlorethamine on weeks 1, 5, and 9; vinblastine and doxorubicin on weeks 1, 3, 5, 7, 9, and 11; etoposide IV over 30-45 minutes for 2 consecutive days on weeks 3, 7, and 11; and vincristine and bleomycin on weeks 2, 4, 6, 8, 10, and 12. Patients also receive oral prednisone every other day on days 1-63 followed by a taper on days 64-84. Treatment continues for 12 weeks.
* Arm II (ABVD): Patients receive doxorubicin, bleomycin, vinblastine, and dacarbazine on days 1 and 15. Treatment repeats every 28 days for 6-8 courses.

All patients achieving a complete remission or partial remission after chemotherapy undergo involved field radiotherapy if they had initial bulky mediastinal disease, initial nodal masses at least 5 cm in diameter, or initial splenic disease.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: Approximately 700-850 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma (any sub-type)

  * Stage IB, IIB, IIIA, IIIB, or IV OR
  * Stage IA or IIA with locally extensive disease (e.g., bulky mediastinal disease (e.g., greater than 0.33 of the maximum transthoracic diameter on routine chest X-ray or at least 2 extranodal sites of disease))

PATIENT CHARACTERISTICS:

Age:

* 18 to 60

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Complete blood count normal unless directly due to Hodgkin's lymphoma

Hepatic:

* Hepatic function normal unless directly due to Hodgkin's lymphoma

Renal:

* Renal function normal unless directly due to Hodgkin's lymphoma

Cardiovascular:

* No pre-existing cardiac disease

Pulmonary:

* No pre-existing pulmonary disease

Other:

* Not pregnant
* Fertile patients must use effective contraception during and for six months after study
* HIV negative
* No other prior malignancy except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior therapy for Hodgkin's lymphoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 850 (Estimated)
Dates: Start 2001-10

PRIMARY OUTCOMES:
Relapse-free survival

SECONDARY OUTCOMES:
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Hoskin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (37):
- United Kingdom (37):
  - Basildon University Hospital, Basildon, England
  - Royal United Hospital, Bath, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Saint Richards Hospital, Chichester, England
  - Walsgrave Hospital, Coventry, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Hemel Hempstead General, Hemel Hempstead, England
  - Hull Royal Infirmary, Hull, England
  - King George Hospital, Ilford, Essex, England
  - Lincoln County Hospital, Lincoln, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - St. George's Hospital, London, England
  - University College Hospital - London, London, England
  - James Paget Hospital, Norfolk, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Oldchurch Hospital, Romford, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - Royal Marsden - Surrey, Sutton, England
  - Torbay Hospital, Torquay, England
  - City Hospital - Birmingham, West Bromwich, England
  - New Cross Hospital, Wolverhampton, England
  - Worthing Hospital, Worthing, England
  - Cancer Care Centre at York Hospital, York, England
  - Craigavon Area Hospital, Craigavon, Northern Ireland
  - Monklands General Hospital, Airdrie, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - South West Wales Cancer Institute, Swansea, Wales